CLINICAL TRIAL: NCT07131150
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of Umbilical Cord Mesenchymal Stem Cell Injection (SC01009) in the Treatment of Idiopathic Pulmonary Fibrosis
Brief Title: Menstrual Blood-Derived Mesenchymal Stem Cell Injection (SC01009) in the Treatment of Idiopathic Pulmonary Fibrosis
Acronym: IPF II
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Jieming QU, Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IPM01-XY1010-2
Record Dates: First submitted 2025-07-14; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Trial Group 1 (Experimental)
  Interventions: Biological: SC01009 injection
- Trial Group2 (Experimental)
  Interventions: Biological: SC01009 injection
- Placebo Group (Placebo Comparator)
  Interventions: Biological: Placebo Group(Vehicle)

INTERVENTIONS:
Biological: SC01009 injection — Menstrual Blood-Derived Mesenchymal Stem Cell (Product Code: SC01009) Injection is a cell therapy product developed by Zhejiang Sinocord Precision Medicine Technology Co., Ltd. The active component consists of mesenchymal stem cells (MSCs) derived from menstrual blood.
  Arms: Trial Group 1; Trial Group2
Biological: Placebo Group(Vehicle) — The placebo consists of the SC01009 Injection formulation solution, containing all components identical to the active product except for the absence of mesenchymal stem cells.
  Arms: Placebo Group

SUMMARY:
At present, the diagnosis of IPF is still difficult and it cannot be completely cured. Treatment is still aimed at improving symptoms and delaying the decline of lung function. The treatment measures for IPF mainly include drug therapy ( pirfenidone and nintedanib), non-drug therapy (such as oxygen therapy, pulmonary rehabilitation), treatment of complications/comorbidities, symptomatic treatment and palliative treatment. However, IPF cannot be completely cured at present, so lung transplantation is a feasible option for the treatment of IPF. However, due to the scarcity of donor lungs, prevention of acute and chronic rejection reactions, post-transplant infection complications, and high costs, its clinical implementation is limited. Therefore, there is still a large unmet treatment need for IPF, and new therapeutic drugs are urgently needed.

In recent years, mesenchymal stem cells (MSCs) have been considered a new hope for the treatment of IPF. MSCs are a type of multipotent stem cells with the potential for self-proliferation and differentiation. They have the characteristics of self-renewal, multidirectional differentiation, low immunogenicity, and paracrine. They can automatically home to damaged areas, promote epithelial tissue repair, inhibit inflammation, and inhibit abnormal proliferation of fibroblasts . Many clinical trials at home and abroad are exploring the effectiveness and safety of MSC in the treatment of pulmonary fibrosis. An Australian study found that in patients with moderate to severe IPF, intravenous infusion of umbilical cord MSCs up to 2 × 106 cells/kg was safe, and no decrease in forced vital capacity (FVC), diffusing vital capacity for carbon monoxide (DLCO), 6-minute walk test distance (6MWD), and CT fibrosis score was observed during a 6-month follow-up . The results of the American AETHER study also showed that a single intravenous infusion of up to 2 × 10^ 8 cells of bone marrow MSCs was safe, with no serious treatment-related adverse events observed. Moreover, 60 weeks after infusion , FVC% decreased by 3.0% and DLCO% decreased by 5.4%, both of which were below the threshold for disease progression .

This study adopted a multicenter, randomized, double-blind, placebo-controlled, parallel design to evaluate the efficacy and safety of SC01009 injection in IPF subjects .

This study plans to enroll 66 subjects, who will be randomly stratified according to whether they have received oral pirfenidone/nintedanib treatment at screening , and randomly assigned to two trial groups and one placebo group in a 1:1:1 ratio.

This study includes a screening period of up to 4 weeks, a 24-week treatment follow-up period, and a 2-year long-term follow-up period. After screening, qualified subjects will be given medication according to the following dosing schedule according to their group:

Trial Group 1: received intravenous infusion of SC01009 injection in week 1, divided into 3 infusions every other day, each infusion of 3 × 10^ 7 cells, with a total dose of 9 × 10 ^7 cells; received intravenous infusion of placebo in week 13, with the same administration method as in week 1; Experimental group 2: received intravenous infusion of SC01009 injection at week 1 and week 13, respectively. Each administration was divided into 3 infusions every other day, with 3 × 10^7 cells in each infusion , and the total dose was 1.8 × 10^8 cells.

Placebo group: received intravenous infusion of placebo at week 1 and week 13, respectively, with the same administration method as the cell therapy group.

After completing 24 weeks of treatment follow-up, all subjects entered the long-term follow-up phase and were unblinded after the study database was locked . The subjects in the original placebo group could end the follow-up, while the subjects receiving cell therapy would continue to be followed up for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily sign the written informed consent (ICF) and agree to complete the trial according to the protocol requirements;
* 2. ≥ 18 and ≤ 80 years old when signing the ICF , regardless of gender;
* 3. Diagnostic Confirmation of IPF;
* 4. ≥ 50% and ≤ 90% at screening ; DLCO% ≥ 30% and ≤ 90% (corrected for hemoglobin [Hb]);
* 5. received nintedanib or pirfenidone treatment for at least 8 weeks before screening and do not plan to start or restart anti-fibrotic treatment; or patients who have received stable nintedanib or pirfenidone treatment for at least 8 weeks before screening and do not receive combination therapy of nintedanib and pirfenidone ;
* 6. 2 ≥ 60 mmHg at screening ; able to complete the 6- minute walk test ( 6MWT ) and walk distance > 150 m;
* 7. are willing to use at least one effective contraceptive method for contraception during the study .

Exclusion Criteria:

* 1. Other lung diseases within 6 months before screening, including chronic obstructive pulmonary disease (forced expiratory volume in 1 second/forced vital capacity (FEV1/FVC) after using bronchodilator < 0.70), emphysema (emphysema occupies ≥ 50% of the entire HRCT according to the central review of HRCT, or the degree of emphysema is greater than the degree of fibrosis), pulmonary hypertension ≥ 50 mmHg indicated by echocardiography , active tuberculosis, pulmonary embolism, uncontrolled asthma, pneumothorax, pneumoconiosis, bronchiolitis obliterans or other active lung diseases;
* 2. In addition to IPF, there are other types of interstitial lung disease (ILD), including ILD with known causes (such as family or occupational environmental exposure, connective tissue disease and drug toxicity, etc.), granulomatous ILD (such as sarcoidosis), and other rare ILD (such as alveolar proteinosis, pulmonary amyloidosis, etc.); among them, for the exclusion of connective tissue disease-related interstitial lung disease ( CTD-ILD), relevant examinations within 12 months before screening were accepted;
* 3. Patients who are in the acute exacerbation stage of IPF at the time of screening, or who have AE-IPF within 3 months before screening (determined by the investigator); AE-IPF is defined as: IPF patients who have a significant acute deterioration of respiratory function in a short period of time, mainly characterized by the new appearance of diffuse ground-glass shadows and/or consolidation shadows in both lungs on the original UIP background on chest HRCT;
* 4. Patients with lung infection or other serious infection requiring intravenous antibiotic treatment within 4 weeks before screening;
* 5. Patients with a history or evidence of major cardiovascular disease within 6 months before screening, including but not limited to: myocardial infarction, coronary angioplasty or bypass surgery, heart valve repair, II or III degree atrioventricular block, malignant arrhythmia ( such as ventricular tachycardia, frequent supraventricular tachycardia, atrial fibrillation, atrial flutter, etc. ), unstable angina, transient ischemic attack, cerebrovascular accident, congestive heart failure with a heart function grade of III or IV of the New York Heart Association (NYHA) , etc.; or left ventricular ejection fraction (LVEF) <50% at screening;
* 6. Patients with a history of tumor (except for patients with cured basal cell carcinoma of the skin, squamous cell carcinoma in situ of the skin, or carcinoma in situ of the cervix), or patients whose tumor marker examinations are determined by the investigator to be clinically significant and may affect safety assessments;
* 7. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 × upper limit of normal (ULN), or total bilirubin (TBIL) >1.5 × ULN at screening;
* 8. Estimated glomerular filtration rate (eGFR) <45 mL/min/1.73m² at screening;
* 9. Patients who are positive for hepatitis B surface antigen (HBsAg) and hepatitis B virus deoxyribonucleic acid (HBV-DNA) ≥ the lower limit of the detection value during screening, or who are positive for hepatitis C virus (HCV) antibody and hepatitis C virus ribonucleic acid (HCV-RNA) ≥ the lower limit of the detection value, or who are positive for human immunodeficiency virus (HIV) antibody, or who are positive for Treponema pallidum antibody (Those who are positive for Treponema pallidum antibody need to undergo non-specific syphilis antibody test and the researchers will determine whether they can participate in the trial);
* 10. Blood pressure is still not controlled after antihypertensive drug treatment within 3 months before screening, and blood pressure during the screening period is ≥ 160/100 mmHg;
* 11. Patients planning to receive lung transplantation or with a history of solid organ transplantation;
* 12. Those who have undergone lung resection; or those who have undergone major surgery (including lung surgery) or unhealed wounds (except for diagnostic surgery or when the investigator determines that the subject has fully recovered from the surgery) within 4 weeks before screening, or those who are planning to undergo major surgery;
* 13. 20 mg/ d (or other glucocorticoids of equivalent dose) within 28 days before screening ;
* 14. Use of cytotoxic drugs (such as chloramphenicol, azathioprine , cyclophosphamide, methotrexate ) or pulmonary hypertension drugs (such as endothelin receptor antagonists [such as bosentan, ambrisentan, macitentan], PDE5 inhibitors [such as sildenafil, tadalafil, vardenafil ]) within 4 weeks or 5 half -lives before screening (whichever is longer) ;
* 15. Use of drugs that may cause pulmonary fibrosis within 6 months before screening, such as amiodarone, bleomycin, etc.;
* 16. Patients who are known or suspected to be allergic to the active or inactive ingredients of the investigational drug (such as dimethyl sulfoxide [DMSO], human serum albumin [HSA], dextran, and compound electrolytes) ;
* 17. Those with a history of drug abuse or other serious mental illness, who may increase the risk of participating in the study or interfere with the study treatment and research results as determined by the researchers;
* 18. Participants who have participated in any other clinical trials within 3 months before screening (except patients who have not received trial drugs); or participated in mesenchymal stem cell clinical trials within 2 years before screening; or received other types of stem cells before screening;
* 19. Other situations that the researcher considers unsuitable for participation in this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in forced vital capacity (FVC) (ml) | Baseline, Week 24

SECONDARY OUTCOMES:
Changes from baseline in the diffusing capacity for carbon monoxide as a percentage of predicted value (DLCO%) | baseline, week 24
a. FVC (ml) decreased by ≥ 10% or DLCO% decreased by ≥ 15% compared with baseline; b. Acute exacerbation of IPF (AE-IPF); c. All-cause mortality occurred; | Time to first clinical worsening event, including any of the following
Changes in FVC (ml) from baseline | weeks 4 and 12
Changes from baseline in forced vital capacity % predicted (FVC%) | weeks 4, 12, and 24 ;
Changes in DLCO% from baseline | weeks 4 and 12
arterial oxygen partial pressure (PaO 2 ) from baseline | weeks 4 , 12 , and 24
Changes from baseline in 6-minute walk test distance (6MWD) | weeks 4, 12, and 24;
Changes from baseline in the Instructions for Completing the Living with Pulmonary Fibrosis Impacts Questionnaire (L-PF Impacts) and Instructions for Completing the Living with Pulmonary Fibrosis Symptoms Questionnaire (L-PF Symptoms) | weeks 4, 12, and 24
  Score range: 0 to 92, higher scores mean a worse outcome
The occurrence of adverse events (AEs)/serious adverse events (SAEs) | Baseline，Day 1 ，up to 24 weeks，2years
  Number of participants with treatment-related adverse events as assessed by CTCAE 5.0，Tumorigenicity assessment during the 2-year observation period following the main observation period
Number of Participants with Post-Treatment Abnormalities in Laboratory tests | Baseline，Day 1， up to 24 weeks
  Number of Participants with Post-Treatment Abnormalities in Laboratory tests (Complete Blood Count, Blood Biochemistry, Urinalysis, Coagulation Function, C-reactive Protein [CRP]) as Assessed by CTCAE v5.0
Number of Participants with Post-Treatment Abnormalities in Vital Signs | Baseline，Day 1 ，up to 24 weeks
  Number of Participants with Post-Treatment Abnormalities in Vital Signs as Assessed by CTCAE v5.0
Number of Participants with post-treatment normality/abnormality transitions | Baseline，Day 1 ，up to 24 weeks
  Number of Participants with post-treatment normality/abnormality transitions (Normal, Abnormal - Not Clinically Significant, Abnormal - Clinically Significant)
12- lead electrocardiogram ( ECG ) examination | Baseline，Day 1， up to 24 weeks
  including heart rate (HR), PR interval , QT interval, RR interval, QTcF and QRS complex duration，Clinical assessment outcomes (Normal, Abnormal - Not Clinically Significant, Abnormal - Clinically Significant) with pre-/post-treatment normality/abnormality transitions
Occurrence of Infusion Reactions | during administration and within 8 hours after completion of administration

OTHER OUTCOMES:
Plasma Drug Concentration of the biomarkers | Week1, 4, 12, 13 , and 24
  the biomarkers（Exploratory Endpoints )

CONTACTS AND LOCATIONS:
Locations (22):
- China (22):
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Chaoyang Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Beijing FriendBeijing Friendship Hospital, Capital Medical UniversityBeijing Friendship Hospital, Capital Medical Universityship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The Second Hospital of Hebei Medical University, Hebei, Hebei
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Union Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Drum Tower Hospital Affiliated to Nanjing University Medical School, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The Second Hospital of Jilin University, Changchun, Jielin
  - Ningxia Medical University General Hospital, Yinchuan, Ningxia
  - Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Air Force Medical University Xijing Hospital, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No